CLINICAL TRIAL: NCT03200340
Title: Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate EC-18 for Oral Mucositis in Patients With Concomitant Chemoirradiation for Cancers of the Mouth, Oropharynx, Hypopharynx and Nasopharynx
Brief Title: EC-18 for Oral Mucositis in Patients With Concomitant Chemoirradiation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: EC-18-202
Record Dates: First submitted 2017-06-13; First posted 2017-06-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Stomatitis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: 2 stages: Stage 1 is a blinded parallel group safety study of 4 cohorts of 24 subjects randomized (1:1:1:1) to receive either EC-18 500 mg, 1000 mg, 2000 mg, or placebo.
  Dosing will commence on the first day of radiation and continue until the last day of radiation. After of 4 weeks, an independent Data Safety Monitoring Board (DSMB) will evaluate safety endpoints in blinded fashion. DSMB assessment will be repeated after completion of dosing. Stage 2 of the study will evaluate both safety and efficacy.
  Eighty (80) subjects will be randomized in a 1:1 scheme to receive placebo or EC-18 at the dose determined in Stage 1. The design of stage 2 is the same as stage 1.
Who Masked: Participant, Investigator
Masking Description: Subjects and investigators will be blinded to treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- [Part 1] Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo
- [Part 1] EC-18 500 mg (Experimental): 1 capsule of EC-18
  Interventions: Drug: EC-18
- [Part 1] EC-18 1000 mg (Experimental): 2 capsules of EC-18 500 mg
  Interventions: Drug: EC-18
- [Part 1] EC-18 2000 mg (Experimental): 4 capsules of EC-18 500 mg
  Interventions: Drug: EC-18
- [Part 2] Placebo (Placebo Comparator): Placebo 2000mg
  Interventions: Drug: Placebo
- [Part 2] EC-18 2000mg (Experimental): RP2D: EC-18 2000mg (Part 1 result)
  Interventions: Drug: EC-18

INTERVENTIONS:
Drug: EC-18 — Oral administration of EC-18 twice daily
  Other Names: EC-18 soft capsules
  Arms: [Part 1] EC-18 1000 mg; [Part 1] EC-18 2000 mg; [Part 1] EC-18 500 mg; [Part 2] EC-18 2000mg
Drug: Placebo — Placebo to match EC-18 capsule administration
  Other Names: Placebo capsule
  Arms: [Part 1] Placebo; [Part 2] Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, 2-stage trial in subjects with squamous cell cancers of the mouth, oropharynx, hypopharynx and nasopharynx planned to receive standard fractionated IMRT-delivered radiotherapy with concomitant chemotherapy (cisplatin). Informed consent will be obtained from each subject prior to enrollment.

The trial will be performed in 2 stages:

Stage 1 will consist of a blinded parallel group safety study of 4 cohorts in which 24 subjects will be randomized (1:1:1:1) into four equally sized groups to receive one of three doses of EC-18 (500 mg, 1000 mg, 2000 mg; unit dose of 500 mg) or placebo. Stage 2 of the study will evaluate both safety and efficacy.

Stage 2 will consist of eighty (80) subjects who will be randomized in a 1:1 scheme to receive either placebo or 2000 mg of EC-18 as determined by iDSMB in Stage 1.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, 2-stage trial in subjects with squamous cell cancers of the mouth, oropharynx, hypopharynx and nasopharynx planned to receive standard fractionated IMRT-delivered radiotherapy with concomitant chemotherapy (cisplatin). Informed consent will be obtained from each subject prior to enrollment.

The trial will be performed in 2 stages:

Stage 1 will consist of a blinded parallel group safety study of 4 cohorts in which 24 subjects will be randomized (1:1:1:1) into four equally sized groups to receive one of three doses of EC-18 (500 mg, 1000 mg, 2000 mg; unit dose of 500 mg) or placebo delivered in the following daily schedule:

TDD AM PM Placebo 2 placebo 2 placebo 500mg 1 active + 1 placebo 2 placebo 1000mg 1 active + 1 placebo 1 active + 1 placebo 2000mg 2 active 2 active Dosing will commence on the first day of radiation (one hour after the first fraction) and continue until the last day of radiation. Test drug will be administered as an oral 500 mg capsule in divided daily doses as indicated above. At the completion of 4 weeks of dosing, an independent Data Safety Monitoring Board (DSMB) will evaluate safety endpoints in blinded fashion. If no safety issues are identified, the DSMB will approve continuation of dosing until the last day of radiation. If a safety issue is noted, the DSMB may unblind the treatment assignment to ascertain if the adverse event is associated with study drug. DSMB assessment will be repeated after completion of dosing (when each subject has been dosed through the last day of radiation). If no safety issues are identified, the efficacy component of the study (Stage 2) will commence using the highest dose of study drug consistent with a positive safety outcome.

Stage 2 of the study will evaluate both safety and efficacy. Eighty (80) subjects will be randomized in a 1:1 scheme to receive either placebo or 2000 mg of EC-18 as determined by iDSMB in Stage 1. Twice daily dosing will begin on the first day of radiation (1 hour after the first fraction) and continue until the last day of radiation (approximately 7 weeks).

The study will be performed in four phases: screening, the active dosing phase, short-term follow-up and long-term follow-up. The screening phase will be performed within 4 weeks of randomization and will determine subjects' eligibility. The active phase will begin on the first day of study drug dosing (also the first day of radiation therapy) and will continue until the last day of radiation therapy. This period typically is 7 weeks depending on the subject's radiation plan. The short-term follow-up phase will begin on the last day of radiation and continue for approximately 4-6 weeks until clinical and symptomatic signs of oral mucositis have resolved. The long-term follow-up phase extends for 12 months following the last dose of radiation and is included to assure that EC-18 does not the impact of tumor response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female age 18 years or older
* Pathologically confirmed diagnosis of squamous cell carcinoma of the mouth, oropharynx, hypopharynx or nasopharynx
* Planned to receive IMRT with daily fractions of 2.0 Gy to 2.2 Gy to a cumulative dose of at least 60 Gy and a maximum of 72 Gy
* Radiation fields to include at least two mucositis sites at risk (buccal mucosa, floor of mouth, ventral and lateral tongue, soft palate) in which both sites receive a minimum cumulative dose of 55 Gy
* Planned to receive concomitant single agent chemotherapy with cisplatin given either weekly or tri-weekly
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Screening Laboratory Values Hemoglobin ≥ 9g/dL White blood cell count ≥ 3,500 cells/mm3 Absolute neutrophil count ≥ 1,500 cells/mm3 Total bilirubin ≤ 2 times upper limit of normal Serum AST and ALT ≤ 2.5 times upper limit of normal Serum creatinine concentration ≤ 2mg/mL Pregnancy test: negative for females of childbearing potential
* Subjects of childbearing potential must consent to utilize a medically accepted means of contraception throughout the active dosing period with study medication and for a minimum of 30 days following the administration of the last dose of study medication.

Exclusion Criteria:

* Unable to provide informed consent or, in the opinion of the Principal Investigator, comply with the protocol.

  * Prior radiation therapy to the head and neck
  * Metastatic disease
  * Presence of active infectious disease excluding oral candidiasis
  * Presence of oral mucositis or any oral lesion that would confound the assessment of oral mucositis
  * Active systemic disease or condition known to impact the risk or course of oral mucositis including chronic immunosuppression and known seropositivity for HIV
  * Use of any investigational agent within 30 days of the first radiation dose
  * Active alcohol abuse syndrome
  * Subjects with a history of hepatitis of any etiology or hepatic insufficiency
  * Pregnant or nursing at the time of signing informed consent
  * Known sensitivity to any study medication
  * Unwilling or unable to complete study diary
  * Any other condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Duration of Severe Oral Mucositis (SOM) during the active treatment and short-term follow-up periods | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Duration of Grade 3 or 4 oral mucositis

SECONDARY OUTCOMES:
Duration of SOM during the active treatment period | 7 Weeks (Active)
  Duration of Grade 3 or 4 oral mucositis
Incidence of severe oral mucositis defined as WHO grade of 3 or 4 during the active treatment period | 7 Weeks (Active)
  Incidence of severe oral mucositis defined as WHO grade of 3 or 4
Incidence of severe oral mucositis defined as WHO grade of 3 or 4 during the active treatment and short-term follow-up periods | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Incidence of severe oral mucositis defined as WHO grade of 3 or 4
Incidence of ulcerative mucositis (defined as WHO grade of 2, 3, or 4) during the active treatment period | 7 Weeks (Active)
  Incidence of WHO grade of 2, 3, or 4 ulcerative mucositis
Incidence of ulcerative mucositis (defined as WHO grade of 2, 3, or 4) during the active treatment and short-term follow-up periods | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Incidence of WHO grade of 2, 3, or 4 ulcerative mucositis
Duration of ulcerative mucositis (WHO criteria) | From the onset to the day when ulcerative mucositis has resolved (up to 22 weeks)
  Duration of grade 3 or 4 ulcerative mucositis
Delay in onset of SOM (WHO criteria) | Start of the radiation treatment (Day 1) until SOM has resolved (up to 22 weeks)
  Time to onset of grade 3 or 4 severe oral mucositis
Reduction in patient-reported mucositis-related mouth pain and analgesic use | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Frequency of disease-related mouth pain and analgesic use

OTHER OUTCOMES:
Duration of severe oral mucositis as defined by RTOG criteria | 7 Weeks
  Duration of severe oral mucositis based on RTOG criteria
Incidence of severe oral mucositis as defined by RTOG criteria | 7 Weeks
  Incidence of severe oral mucositis as defined by RTOG criteria
Duration of severe oral mucositis as defined by NCI-CTCAE v.4 criteria | 7 Weeks
  Duration of severe oral mucositis based on NCI-CTCAE v.4 criteria
Incidence of severe oral mucositis as defined by NCI-CTCAE v.4 criteria | 7 Weeks
  Incidence of severe oral mucositis based on NCI-CTCAE v.4 criteria
Patient reported outcomes as measured by the Oral Mucositis Daily Questionnaire (OMDQ) | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Patient reported outcomes based on 0-4 and 0-10 scales (measuring quality of life)
Patient reported outcomes as measured by Weekly Functional Assessment of Cancer Therapy-for Patients with Head & Neck Cancer (FACT-HN) | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Patient reported outcomes based on 0-4 scale (measuring quality of life)
Breaks in radiation delivery | 7 Weeks
  Frequency of interruptions in radiation therapy
Break duration in radiation delivery | 7 Weeks
  Duration of interruptions in radiation therapy
Healthcare resource use including reliance on gastrostomy feeding, unplanned office visits, emergency room visits, and hospitalizations | 7 Weeks (Active) + 4-6 Weeks (STFU)
  Number of subjects who utilized healthcare resources listed above

CONTACTS AND LOCATIONS:
Overall Officials: Dong Moon Shin, MD, Principal Investigator — Emory University Winship Cancer Institute; Mahesh Kudrimoti, MD, Principal Investigator — University of Kentucky, Chandler Medical Center, CCTS
Locations (20):
- United States (20):
  - Veterans Affairs Long Beach Health Care System, Long Beach, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Kentucky, Chandler Medical Center, CCTS, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai - Union Square, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - VA Portland HealthCare System, Portland, Oregon
  - St. Luke's Cancer Center - Anderson Campus, Easton, Pennsylvania
  - Hope Cancer Center of East Texas, Tyler, Texas
  - Baylor Scott & White Medical Center - Hillcrest, Waco, Texas
  - MultiCare Institute for Research and Innovation, Spokane, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No